CLINICAL TRIAL: NCT06175585
Title: Construction of a Theoretical Model of Medical Behavior of Patients With Chronic Kidney Disease From the Perspective of Supply: An Empirical Analysis Based on Andersen Behavior Model
Brief Title: Construction of Theoretical Model of Medical Treatment Behavior of Patients With Chronic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Zheng Jie, Associate professor, Shanxi Medical University
Other Study IDs: 2019041044-1
Record Dates: First submitted 2023-12-04; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Narrative Nursing; Maintenance Hemodialysis; Chronic Kidney Diseases
Keywords: self-efficacy; negative emotions; life quality
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- traditional nursing group
  Interventions: Other: traditional nursing
- narrative nursing group
  Interventions: Other: narrative nursing

INTERVENTIONS:
Other: narrative nursing — The narrative nursing process is based on the practice of "two-line system" proposed by Jiang, which is carried out in a separate classroom, office or ward with sufficient space and good lighting. The environment is set to the right temperature and humidity for comfortable face-to-face conversation. This process is done in stages, depending on how often the patient is dialysis three or more times a week.
  Each session lasts about 30 minutes and the whole process lasts four weeks. Adjust to the specific needs of each patient .
  Groups: narrative nursing group
Other: traditional nursing — Patients undergoing MHD received traditional nursing interventions, encompassing various aspects such as dietary advice, instructions on medication usage, health education, emphasis on precautions during dialysis, and guidelines for vascular access care. Additionally, the nurses proactively inquired about patients' emotional well-being during the nursing shift change, actively engaged and uplifted patients experiencing low spirits, and encouraged family members to provide emotional support.
  Groups: traditional nursing group

SUMMARY:
The impact of narrative nursing interventions on negative emotions, self-efficacy, quality of life in individuals undergoing maintenance hemodialysis

DETAILED DESCRIPTION:
The objective of this study is to create a narrative nursing protocol using the "two-line system" approach to enhance the practice of narrative nursing.Investigators applied this protocol during maintenance hemodialysis (MHD) treatment, with the aim of examining the impact of the interventions on negative emotions, self-efficacy, and overall quality of life of patients. By analyzing the data before and after the interventions, investigators aim to demonstrate how targeted narrative nursing measures can positively influence negative emotions, self-efficacy, and life quality of patients.

ELIGIBILITY:
Inclusion criteria:

* Patients diagnosed with ESRD and treated with dialysis for more than 3 months;
* Patients aged ≥18 years old;
* Patients with complete clinical data;
* Patients who are clearly conscious and can accurately express their willingness;
* Patients who have signed informed consent and are willing to cooperate with the study.

Exclusion criteria:

* Patients with other serious systemic diseases, such as severe cardiovascular and cerebrovascular diseases, severe diabetes, etc.;
* Patients with mental disorder, such as cognitive or intellectual disability;
* Patients with a history of anxiety and depression;
* Patients with intermittent loss of consciousness or are unable to understand the questions in the questionnaire.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing MHD at the Department of Nephrology in our hospital.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2024-11-29 (Estimated); Study Completion 2024-12-29 (Estimated)

PRIMARY OUTCOMES:
Zung's Self-Rating Anxiety Scale | one week
  assess the anxiety and depression levels of patients
Self-rating Depression Scale | one week
  assess the anxiety and depression levels of patients

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: Yes